CLINICAL TRIAL: NCT07346820
Title: VDJ-recombination of the B-cell Receptor Following Hematopoietic Stem Cell Transplantation, an Observational Study
Brief Title: VDJ-recombination of the B-cell Receptor Following Hematopoietic Stem Cell Transplantation
Acronym: VReST
Status: Not yet recruiting | Type: Observational
Sponsor: Umeå University (Other)
Collaborators: Region Västerbotten (Other Government)
Responsible Party: Sponsor
Other Study IDs: The VReST study
Record Dates: First submitted 2025-12-19; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Stem Cell Transplantation, Hematopoietic; V(D)J Recombination; Receptors, Antigen, B-Cel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients undergoing autologous stem cell transplantation
- Patients undergoing allogenic stem cell transplantation
- Stem cell donors

SUMMARY:
When a person undergoes a stem cell transplant-an important procedure used to treat serious blood diseases such as leukaemia, lymphoma, or myeloma-the entire immune system is affected. The transplant essentially "resets" the immune system, meaning that the patient loses much of the protection against infections that has been built up over a lifetime. After the transplant, the patient therefore needs to be revaccinated against several diseases, such as tetanus, diphtheria, polio, COVID-19, and pneumococcal disease.

In this study, we aim to investigate how B cells-the immune cells that produce antibodies-reconstitute after a stem cell transplant. We are particularly interested in a genetic process called VDJ recombination, through which each B cell develops a unique receptor that enables it to recognize and fight a specific virus or bacterium. This process is what makes our immune system so effective. But what happens to this diversity after the entire immune system has been restarted with new stem cells? Does the body regain the same ability to recognize pathogens? Are there differences between patients who receive their own stem cells (autologous transplantation) and those who receive stem cells from another person (allogeneic transplantation)?

To answer these questions, we will follow patients undergoing stem cell transplantation at Umeå University Hospital. We will collect blood samples before and after the transplantation and will assess whether-and how well-patients generate antibodies in response to the vaccines given after transplantation. Using flow cytometry and genetic analyses, we will examine both which B-cell populations are generated and what their genetic architecture looks like. The goal is to understand how the new immune system is rebuilt after transplantation and, ultimately, to help improve vaccination strategies and infection prevention for this vulnerable patient group

DETAILED DESCRIPTION:
Purpose and aims

The humoral immune system is critical for mounting protective responses against severe microbial infections. This is a highly specific response, where naïve B cell clones that recognize epitopes on a pathogen are activated, clonally expands and differentiates to memory B cells and antibody producing plasma cells.

The specificity of the response is dependent on VDJ recombination that creates naïve B cell clones, each with a distinct B cell receptor that carry unique variable (V), diversity (D) and joining segments. While the process of VDJ recombination is well investigated, it is not well established how/if VDJ recombination is affected in B cells after autologous or allogeneic stem cell transplantation. Such knowledge may improve on strategies to re-vaccinate vulnerable patient groups that require stem cell transplantation to alleviate a number of haematological disorders. Here, we will utilize samples from individuals before and after haematological stem cell transplantation to better define the impact on VDJ recombination and clonal responses to vaccine antigens.

Background

Stem cell transplantation is a procedure where most/all hematopoietic cells are eradicated from a patient and replaced by new stem cells that are derived from "self" (autologous) or from an MHC matched donor. Upon a successful stem cell transfer, new and healthy hematopoietic cells will emerge. After the procedure immunity to several vaccine preventable diseases are lost or severely impaired putting the patient at risk.

Following transplantation patients are vaccinated against several infectious diseases according to an established vaccine schedule. This provides an opportunity to study VDJ recombination in a situation where the immune system is "reset" - compare and contrast the situation to before the procedure as well as differences between autologous and allogenic transplantation.

A standardized vaccination schedule based on recommendations by the European Conference on Infections in Leukemia (ECIL) is implemented to HSCT patients. Vaccinations against pneumococcal infections, capsulated haemophilus influenzae, tetanus, diphtheria, polio, pertussis, covid19 and influenzae are recommended to all. Further vaccination may be considered according to the preferences of the patient.

B cells are critical for humoral immune responses, as they specifically respond to an antigen and then differentiate into antibody producing plasma cells, and to memory B cells. The importance of this for protection against a primary infection is readily illuminated by susceptibility to severe infectious disease if the humoral immune system is defect or after treatment with B cell depleting drugs, such as anti-CD20 antibodies. In addition, the generation of immunological memory then protects us against re-infection with the same pathogen. Of critical importance for this response is the antigen-specificity of the B-cell receptor (BCR) of naïve B cell clones.

The BCR comprise an immunoglobin heavy and light chain with a distinct specificity. The specificity is created by VDJ recombination where one of numerous V, D and J segments are combined into a VDJ region of the heavy chain, and one of numerous V and J segments are combined into a light chain. The combination of these ensures that emerging naïve B cell clones each has a distinct and unique capacity to recognize an epitope. The diversity that is generated ensures that the immune system can respond clonally to almost any foreign pathogen it encounters. By BCR sequencing of B cells, it is therefore possible to determine exactly which V, D or J segments has randomly been recombined to recognize a specific antigen. T cells undergo a similar process of VDJ recombination after maturation in the thymus.

After stem cell transplantation, the VJ-segment of the beta chain T cell receptor develop with a relative symmetry but reduced complexity, as compared with the donor. This may explain why B cells may demonstrate reduced T cell-dependent somatic hypermutation after transplantation. However, it is not well understood if a similar set of B cell clones will emerge after autologous stem cell transplantation or that of an allogenic donor. Since stem cell transplant patients undergo vaccination, this will allow us to closely study the process of antigen-specific VDJ recombination pre- and post "reset" of the immune system, and to couple this to antigenspecific responses after vaccination. We hypothesize that this will reveal further information of how/if the nature of the transplant will affect downstream VDJ recombination and lead to an altered capacity or pattern of immune recognition.

Moreover, it has been shown that impaired humoral immune responses during ageing may be dependent on extrinsic rather that intrinsic factors that affect Bcl6 and CD39-expression the T cell compartment. The potential availability of samples from allogenic donors with age variation will allow for potential verification of these results in humans.

Project description

Study structure

This is an observational cohort study following patients after stem cell transplantation examining the B-cell development following the standardized and established vaccine schedule given as part of clinical practice. In the current version of this schedule in Västerbotten vaccinations against pneumococci, haemophilus influenzae, COVID-19, tetanus, diphtheria, polio and whopping cough are included. Measles, mumps and rubella vaccination may be given following negative immunity test at 24 months from transplantation.

Sampling

i. Sampling before immunosuppressive medication is initiated

ii. Sampling when admitted for stem cell transplantation

iii. Sampling prior to each vaccination time point up until 24 months from transplantation.

iv. In allogenic transplantation sampling of related donor if available (sampling once).

Blood sample analysis

B cell characterization and VDJ sequencing

Antigen specific identification of B cells; We will use established methodology to detect antigen specific B cells. In brief, biotin- and fluorochrome labelled SARS-CoV-2 protein or Influenza type A hemagglutinin protein will be utilized to determine vaccine specific CD19+ CD20+ B cells by flow cytometry. We will focus on cells that has undergone thymus-dependent B cell responses (CD27+IgD-) and phenotype these for activation markers such as DAF and CD71.

For examination of the VDJ repertoire preand post transplantation, we will mainly rely on bulk sequencing but may subject samples to single cell sequencing to reveal if heavy and light chain pairing is affected by the transplantation. We also aim to dissect transcriptional patterns in B cells to reveal specific patterns or molecules that actively predict efficient establishment of Bmem or plasmablasts after stem cell transplantation. For transcriptional patterns, we will perform 10x Chromium single cell gene expression to provide the single cell transcriptome from up to 10,000 vaccine-specific Bmem cells. By combinatorial analysis of both phenotypic and transcriptomic data, we will be able to identify biomarkers or gene expression patterns that predict robust establishment of "boostable" immune memory after stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Willing and able to participate in all parts of the study.
* Signed written consent.
* Patients with a plasma cell disease of lymphoma that qualify for autologous hematological stem cell transplantation determined by the attending physician OR Patients with a condition for which allogenic stem cell transplantation could be needed and qualify for haematological stem cell transplantation according to the attending physician OR Stem cell donor, donating to a study participant.

Exclusion Criteria:

* Unable to give informed consent.
* Not suitable for participation in the study according to the view of the attending physician.
* Previous participation in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who fulfill the inclusion criteria and will receive their stem cell transplantation at the department of hematology at the Umeå university hospital
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2036-12-31 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
VDJ recombination of the B-cell receptor (BCR) after autologous and allogenic stem cell transplantation compared to samples from before transplantation or to samples from stem cell donor. For comparison IgM and IgG antibody levels will also be measured. | From inclusion until end of study which is 24 months after transplantation
  The study will examine the BCR development and VDJ recombination after stem cell transplantation in response to exposure to different vaccine antigens compared to the samples taken before transplantation or samples from the stem cell donor when available. Because the lack of previous studies and by being an exploratory study it is not possible to define quantitative measurable endpoints.
Differences in response to vaccine antigens following autologous stem cell transplantation compared to allogenic stem cell transplantation in VDJ recombination of the B-cell receptor and in IgM and IgG antibody levels. | From inclusion until end of study which is 24 months after transplantation
  The study will examine the BCR development and VDJ recombination after stem cell transplantation in response to exposure to vaccine antigens compared to the before transplantation or to the stem cell donor. Because the lack of previous studies and by being an exploratory study it is not possible to define quantitative measurable endpoints..

CONTACTS AND LOCATIONS:
Locations (1):
- Umeå university hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the sensitive nature of the clinical and biological data collected in this observational study.

REFERENCES:
- [Background] Sorror ML, Maris MB, Storb R, Baron F, Sandmaier BM, Maloney DG, Storer B. Hematopoietic cell transplantation (HCT)-specific comorbidity index: a new tool for risk assessment before allogeneic HCT. Blood. 2005 Oct 15;106(8):2912-9. doi: 10.1182/blood-2005-05-2004. Epub 2005 Jun 30. PMID 15994282
- [Background] Dernstedt A, Leidig J, Holm A, Kerkman PF, Mjosberg J, Ahlm C, Henriksson J, Hultdin M, Forsell MNE. Regulation of Decay Accelerating Factor Primes Human Germinal Center B Cells for Phagocytosis. Front Immunol. 2021 Jan 5;11:599647. doi: 10.3389/fimmu.2020.599647. eCollection 2020. PMID 33469456
- [Background] Kaku CI, Champney ER, Normark J, Garcia M, Johnson CE, Ahlm C, Christ W, Sakharkar M, Ackerman ME, Klingstrom J, Forsell MNE, Walker LM. Broad anti-SARS-CoV-2 antibody immunity induced by heterologous ChAdOx1/mRNA-1273 vaccination. Science. 2022 Mar 4;375(6584):1041-1047. doi: 10.1126/science.abn2688. Epub 2022 Feb 10. PMID 35143256
- [Background] Fisher JS, Adan-Barrientos I, Kumar NR, Lancaster JN. The aged microenvironment impairs BCL6 and CD40L induction in CD4+ T follicular helper cell differentiation. Aging Cell. 2024 Jun;23(6):e14140. doi: 10.1111/acel.14140. Epub 2024 Mar 13. PMID 38481058
- [Background] Suzuki I, Milner EC, Glas AM, Hufnagle WO, Rao SP, Pfister L, Nottenburg C. Immunoglobulin heavy chain variable region gene usage in bone marrow transplant recipients: lack of somatic mutation indicates a maturational arrest. Blood. 1996 Mar 1;87(5):1873-80. PMID 8634435
- [Background] Meier JA, Haque M, Fawaz M, Abdeen H, Coffey D, Towlerton A, Abdeen A, Toor A, Warren E, Reed J, Kanakry CG, Keating A, Luznik L, Toor AA. T Cell Repertoire Evolution after Allogeneic Bone Marrow Transplantation: An Organizational Perspective. Biol Blood Marrow Transplant. 2019 May;25(5):868-882. doi: 10.1016/j.bbmt.2019.01.021. Epub 2019 Jan 21. PMID 30677510
- [Background] Cesaro S, Mikulska M, Hirsch HH, Styczynski J, Meylan S, Cordonnier C, Navarro D, von Lilienfeld-Toal M, Mehra V, Marchesi F, Besson C, Masculano RC, Beutel G, Einsele H, Maertens J, de la Camara R; ECIL 9; Ljungman P, Pagano L. Update of recommendations for the management of COVID-19 in patients with haematological malignancies, haematopoietic cell transplantation and CAR T therapy, from the 2022 European Conference on Infections in Leukaemia (ECIL 9). Leukemia. 2023 Sep;37(9):1933-1938. doi: 10.1038/s41375-023-01938-5. Epub 2023 Jul 17. No abstract available. PMID 37460673
- [Background] Cordonnier C, Einarsdottir S, Cesaro S, Di Blasi R, Mikulska M, Rieger C, de Lavallade H, Gallo G, Lehrnbecher T, Engelhard D, Ljungman P; European Conference on Infections in Leukaemia group. Vaccination of haemopoietic stem cell transplant recipients: guidelines of the 2017 European Conference on Infections in Leukaemia (ECIL 7). Lancet Infect Dis. 2019 Jun;19(6):e200-e212. doi: 10.1016/S1473-3099(18)30600-5. Epub 2019 Feb 8. PMID 30744963
- See also: Vaccination schedule after stem cell transplantation used in Umeå — https://rvlitablobprod.blob.core.windows.net/rvlitablobprod/73697.pdf